CLINICAL TRIAL: NCT02680587
Title: Phase II Randomized Observation Versus Stereotactic Ablative RadiatIOn for OLigometastatic Prostate CancEr (ORIOLE) Trial
Brief Title: Stereotactic Body Radiation for Prostate Oligometastases
Acronym: ORIOLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J15180; IRB00079078 (Other: JHMIRB)
Record Dates: First submitted 2016-02-08; First posted 2016-02-11 (Estimated); Results first posted 2021-12-22 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer; Oligometastases
Keywords: Prostate Cancer; Stereotactic Body Radiation Therapy; Stereotactic Ablative Radiotherapy; Oligometastasis
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observational (no SBRT) (No Intervention): Men with oligometastatic prostate cancer lesions randomized to observation
- SBRT (Experimental): Men with oligometastatic prostate cancer lesions randomized to stereotactic body radiation therapy (SBRT).
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — SBRT (1-5 fractions) will be administered.
  Other Names: Stereotactic Body Radiation; Stereotactic Ablative Radiotherapy
  Arms: SBRT

SUMMARY:
Men with oligometastatic prostate cancer lesions will be randomized (1:2) to observation versus SBRT. The study will NOT be blinded. Within three weeks of the initial treatment planning, SBRT (1-5 fractions) will be administered.

DETAILED DESCRIPTION:
This research is being done to determine if we can improve the outcome of prostate cancer patients who have failed primary treatment - surgery or local radiation to the prostate - and have 3 or fewer bone metastases. Patients with metastatic prostate cancer disease will usually be placed on hormonal therapy which can work well for a period of time, but hormonal therapy can have side effects that greatly trouble men. Any effort to delay the start of hormonal therapy would be an advantage to the patient. Radiation treatment usually takes many weeks to deliver and is not given in a high enough doses to metastases to prevent them from coming back locally. Stereotactic body radiation therapy (SBRT) is highly focused radiation, given in a very dose intensive fashion and delivered in usually less than one week. Stereotactic body radiation has been shown to be very effective on bone metastases. Therefore, we are studying the effects of stereotactic body radiation treatment on patients with five or fewer prostate cancer bone metastases to determine if we can stall the use of hormonal therapy and/or prevent other bone metastases from developing elsewhere in the body.

Additionally, fundamental analysis of the oligometastatic state with be achieved through correlation with investigational DCFPyL-positron emission tomography (PET) imaging, which can help us find cancer that has spread (metastatic disease) from its original site in people who have cancer in their prostate to other parts of their body.

Specifically, 54 men with biochemically recurrent, oligometastatic prostate adenocarcinoma will be accrued across 3 centers in the United States. Patients were stratified by primary intervention (surgery vs radiotherapy), prior hormonal therapy, and PSA doubling time, then randomized 2:1 to SBRT or observation. The primary clinical endpoint is progression at 6 months from randomization with the hypothesis that SBRT to all metastases will forestall progression by disrupting the metastatic process. Secondary clinical endpoints include local control at 6 months post-SBRT, SBRT-associated toxicity and quality of life, and ADT-free survival (ADT-FS).

Alterations in the biology of the oligometastatic state induced by stereotactic ablative radiotherapy (SABR) will be investigated using leading-edge correlatives, including: analysis of circulating tumor cells (CTCs; Epic Sciences, San Diego, CA), deep sequencing of circulating tumor DNA (ctDNA) using Cancer Personalized Profiling by deep sequencing (CAPP-Seq) to non-invasively assess tumor burden, and ImmunoSEQ profiling of T-cell repertoires to elucidate the immunological response to SABR (Adaptive Technologies, Seattle, WA). Lastly, the use of the Color Genomics platform (Burlingame, CA), a hereditary cancer assay assessing pathogenic mutations in 30 cancer predisposition genes that account for >90% of the germline mutations known to occur in men with castrate resistant metastatic prostate cancer (mCRPC), will help inform and allow for efforts to advance a more personalized medicine approach to tailor screening and therapies in these men.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have at least one and up to three asymptomatic metastatic tumor(s) of the bone or soft tissue develop within the past 6-months that are ≤ 5.0 cm or <250 cm3.
* Patient must have had their primary tumor treated with surgery and/or radiation.
* Histologic confirmation of malignancy (primary or metastatic tumor).
* PSADT <15 months. PSA doubling time (PSADT) will be calculated using as many PSA values that are available from time of relapse (PSA > 0.2). To calculate PSADT, the Memorial Sloan Kettering Cancer Center Prostate Cancer

Prediction Tool will be used. It can be found at the following web site:

https://www.mskcc.org/nomograms/prostate/psa-doubling-time.

* Patient may have had prior systemic therapy and/or ADT associated with treatment of their primary prostate cancer. Patient may have had ADT associated with salvage radiation therapy (to the primary prostate cancer or pelvis is allowed).
* PSA >1 but <50.
* Testosterone > 125 ng/dL.
* Patient must have a life expectancy ≥ 12 months.
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Patient must have normal organ and marrow function as defined as:

Leukocytes >2,000/μL Absolute Neutrophil Count >1,000/μL Platelets >50,000/μL

- Patient must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* No more than 3 years of ADT is allowed, with the most recent ADT treatment having occurred greater than 6 months prior to enrollment.
* DCFPyL-PET/MRI or DCFPyL-PET/CT scan within the past 6 months with results that demonstrate more disease lesions than baseline CT/Bone Scan
* Castration-resistant prostate cancer (CRPC).
* Suspected pulmonary and/or liver metastases (greater >10 mm in largest axis).
* Patient receiving any other investigational agents.
* Patient is participating in a concurrent treatment protocol.
* Total bilirubin > 3 times the upper limit of normal.
* Liver Transaminases > 5-times the upper limit of normal.
* Unable to lie flat during or tolerate PET/MRI, PET/CT or SBRT.
* Liver Transaminases > 5-times the upper limit of normal.
* Prior salvage treatment to the primary prostate cancer or pelvis is allowed.
* Refusal to sign informed consent.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phuoc Tran, M.D., Principal Investigator — Johns Hopkins Department of Radiation Oncology and Molecular Radiation Sciences
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phillips R, Shi WY, Deek M, Radwan N, Lim SJ, Antonarakis ES, Rowe SP, Ross AE, Gorin MA, Deville C, Greco SC, Wang H, Denmeade SR, Paller CJ, Dipasquale S, DeWeese TL, Song DY, Wang H, Carducci MA, Pienta KJ, Pomper MG, Dicker AP, Eisenberger MA, Alizadeh AA, Diehn M, Tran PT. Outcomes of Observation vs Stereotactic Ablative Radiation for Oligometastatic Prostate Cancer: The ORIOLE Phase 2 Randomized Clinical Trial. JAMA Oncol. 2020 May 1;6(5):650-659. doi: 10.1001/jamaoncol.2020.0147. PMID 32215577
- [Background] Radwan N, Phillips R, Ross A, Rowe SP, Gorin MA, Antonarakis ES, Deville C, Greco S, Denmeade S, Paller C, Song DY, Diehn M, Wang H, Carducci M, Pienta KJ, Pomper MG, DeWeese TL, Dicker A, Eisenberger M, Tran PT. A phase II randomized trial of Observation versus stereotactic ablative RadiatIon for OLigometastatic prostate CancEr (ORIOLE). BMC Cancer. 2017 Jun 29;17(1):453. doi: 10.1186/s12885-017-3455-6. PMID 28662647
- [Derived] Marvaso G, Corrao G, Zaffaroni M, Vincini MG, Lorubbio C, Gandini S, Fodor C, Netti S, Zerini D, Luzzago S, Mistretta FA, Venetis K, Cursano G, Burla T, Mazzocco K, Cattani F, Petralia G, Fusco N, Pravettoni G, Musi G, De Cobelli O, Tang C, Ost P, Palma DA, Orecchia R, Jereczek-Fossa BA. ADT with SBRT versus SBRT alone for hormone-sensitive oligorecurrent prostate cancer (RADIOSA): a randomised, open-label, phase 2 clinical trial. Lancet Oncol. 2025 Mar;26(3):300-311. doi: 10.1016/S1470-2045(24)00730-7. PMID 40049196
- [Derived] Deek MP, Van der Eecken K, Sutera P, Deek RA, Fonteyne V, Mendes AA, Decaestecker K, Kiess AP, Lumen N, Phillips R, De Bruycker A, Mishra M, Rana Z, Molitoris J, Lambert B, Delrue L, Wang H, Lowe K, Verbeke S, Van Dorpe J, Bultijnck R, Villeirs G, De Man K, Ameye F, Song DY, DeWeese T, Paller CJ, Feng FY, Wyatt A, Pienta KJ, Diehn M, Bentzen SM, Joniau S, Vanhaverbeke F, De Meerleer G, Antonarakis ES, Lotan TL, Berlin A, Siva S, Ost P, Tran PT. Long-Term Outcomes and Genetic Predictors of Response to Metastasis-Directed Therapy Versus Observation in Oligometastatic Prostate Cancer: Analysis of STOMP and ORIOLE Trials. J Clin Oncol. 2022 Oct 10;40(29):3377-3382. doi: 10.1200/JCO.22.00644. Epub 2022 Aug 24. PMID 36001857
- See also: Gleason Score Description — https://www.cancer.gov/publications/dictionaries/cancer-terms/def/gleason-score

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 26 Excluded from 80, these are: 19 Did not meet inclusion criteria; 5 Declined to participate; 2 Insurance denied
Groups:
- Observational (no SBRT): Evaluating men with oligometastatic prostate cancer lesions randomized to observation
  Observational (no SBRT): These patient will not receive SBRT. They will be observed.
- SBRT: Evaluating men with oligometastatic prostate cancer lesions randomized to stereotactic body radiation therapy (SBRT).
  SBRT: SBRT (1-5 fractions) will be administered.
Period: Overall Study
Arm/Group | Observational (no SBRT) | SBRT
Started | 18 | 36
Completed | 17 | 36
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Observational (no SBRT): Evaluating males with oligometastatic prostate cancer lesions randomized to observation
  Observational (no SBRT): These patients will not receive SBRT. They will be observed.
- SBRT: Evaluating males with oligometastatic prostate cancer lesions randomized to stereotactic body radiation therapy (SBRT).
  SBRT: SBRT (1-5 fractions) will be administered.
- Total: Total of all reporting groups
Arm/Group | Observational (no SBRT) | SBRT | Total
Number analyzed (Participants) | 18 | 36 | 54
Age, Continuous [Median (Full Range); unit: Years] | 68 [64 to 76] | 68 [61 to 70] | 68 [61 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 36 | 54
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 36 | 54
Initial T stage (extent of the tumor) [Count of Participants; unit: Participants] — Staging for prostate cancer is determined by the American Joint Committee on Cancer guidelines in place at the time of the initial diagnosis/treatment (prior to entry on the study). T-staging is used for tumor size TX: Main tumor cannot be measured. T0: Main tumor cannot be found. T1, T2, T3, T4: Refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues.
  Participants
    cT1c | 1 | 3 | 4
    cT2a | 0 | 2 | 2
    cT2b | 1 | 0 | 1
    cT3a | 1 | 1 | 2
    pT2 | 6 | 12 | 18
    pT3a | 8 | 10 | 18
    pT3b | 1 | 8 | 9
Initial N stage (extent of spread to the lymph nodes [Count of Participants; unit: Participants] — Staging for prostate cancer is determined by the American Joint Committee on Cancer guidelines in place at the time of the initial diagnosis/treatment (prior to entry on the study). N-staging is used in classifying the extent of spread to lymph nodes.
  NX: Cancer in nearby lymph nodes cannot be measured. N0: There is no cancer in nearby lymph nodes. N1, N2, N3: Refers to the number and location of lymph nodes that contain cancer. The higher the number after the N, the more lymph nodes that contain cancer.
  Participants
    N0 | 16 | 31 | 47
    N1 | 1 | 2 | 3
    NX | 1 | 3 | 4
Tumor margin status [Count of Participants; unit: Participants] — Evaluated only among patients with surgery. Patients with radiotherapy are not applicable for this. The tumor margin status following treatment is described by the residual tumor (R) classification: R0, no residual tumor; R1, microscopic residual tumor; R2, macroscopic residual tumor. Residual tumor may be found in the area of primary tumor and its regional lymph nodes and/or at distant sites.
  Participants
    R0 | 10 | 20 | 30
    R1 | 5 | 10 | 15
    Not applicable | 3 | 6 | 9
Gleason score [Count of Participants; unit: Participants] — "A way of describing prostate cancer based on how abnormal the cancer cells in a biopsy sample look under a microscope and how quickly they are likely to grow and spread. Gleason score is calculated by adding together the two grades of cancer cells that make up the largest areas of the biopsied tissue sample. The Gleason score usually ranges from 6 to 10. The lower the Gleason score, the more the cancer cells look like normal cells and are likely to grow and spread slowly".
  Participants
    3+3=6 | 0 | 3 | 3
    3+4=7 | 4 | 8 | 12
    4+3=7 | 4 | 14 | 18
    4+4=8 | 1 | 4 | 5
    4+5=9 | 8 | 4 | 12
    5+4=9 | 0 | 3 | 3
    5+5=10 | 1 | 0 | 1
Initial management [Count of Participants; unit: Participants]
  Surgery | 15 | 30 | 45
  Radiotherapy | 3 | 6 | 9
Time to first recurrence [Median (Full Range); unit: month] | 22 [9 to 51] | 22 [9 to 42] | 22 [9 to 51]
Had received prior ADT [Count of Participants; unit: Participants] | 5 | 28 | 33
Baseline prostate-specific antigen (PSA) [Median (Full Range); unit: ng/dl] | 7 [3 to 17] | 6 [2 to 13] | 6 [2 to 17]
Baseline prostate-specific antigen doubling time (PSADT) [Median (Full Range); unit: months] | 6 [4 to 11] | 8 [4 to 11] | 8 [4 to 11]

OUTCOME MEASURES:

1. Primary Outcome: Progression at 6 Months
Description: Number of participants who progressed at 6 months. Progression is defined as either: 1) a ≥ 25% increase in PSA from nadir (and by ≥ 2 ng/mL), requiring confirmation ≥ 4 weeks later (PCWG2 criteria); and/or, 2) clinical/radiographic-progression defined as symptomatic progression (worsening disease-related symptoms or new cancer-related complications), or radiologic progression (on CT scan: ≥ 20% enlargement in sum diameter of soft-tissue target lesions [RECIST1.1 criteria]; on bone scan: ≥ 1 new bone lesions),initiation of ADT or death due to any cause, whichever occurs first.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Observational (no SBRT) | SBRT
Number analyzed (Participants) | 18 | 36
Participants | 11 | 7

2. Secondary Outcome: Time to Local Progression
Description: Number of months until local progression in patients with oligometastatic disease.
Time Frame: up to 6 months
Measure: Median (Full Range); unit: Months
Arm/Group | Observational (no SBRT) | SBRT
Number analyzed (Participants) | 18 | 36
Months | 5.8 [1 to 6] | 6 [3 to 6]

3. Secondary Outcome: Local Control of SBRT Group
Description: Number of lesions that did not increase in size by at least 20% or more on CT from baseline to 6 months.
Time Frame: 6 months
Population: Data for this outcome measure was not collected from the Observation arm.
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Observational (no SBRT) | SBRT
Number analyzed (Participants) | 0 | 36
Number analyzed (lesions) | 0 | 89
lesions |  | 89

4. Secondary Outcome: Toxicity as Assessed by Number of Participants With Adverse Events Grade 3 or Higher
Description: Number of participants experiencing adverse events Grade 3 or higher, as defined by CTCAE.
Time Frame: up to 6 months
Measure: Number; unit: participants
Arm/Group | Observational (no SBRT) | SBRT
Number analyzed (Participants) | 18 | 36
participants
  3 months | 0 | 0
  6 months | 0 | 0

5. Secondary Outcome: Toxicity as Assessed by Number of Participants With Adverse Events Grades 1 or 2
Description: Number of participants experiencing adverse events Grades 1 or 2, as defined by CTCAE
Time Frame: up to 6 months
Population: 2 from observation group discontinued intervention because of progression prior to 90 days.
Measure: Number; unit: participants
Arm/Group | Observational (no SBRT) | SBRT
Number analyzed (Participants) | 16 | 36
participants
  3 month | 11 | 30
  6 month | 3 | 15

6. Secondary Outcome: Change in Quality of Life as Assessed by Brief Pain Inventory
Description: We will assess quality of life following completion of Stereotactic Body Radiation Therapy via Brief Pain Inventory questionnaire made up of 9 questions. Each question scores from 0-10, with higher scores mean worse outcome or more pain. An overall score, calculated by adding the scores for questions 2, 3, 4 and 5 and then dividing by 4, will be calculated pre-treatment and at the time of day 180. The change in score (between baseline and 6 months) will be evaluated.
Time Frame: Baseline and 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Observational (no SBRT) | SBRT
Number analyzed (Participants) | 18 | 36
score on a scale | 0 [0 to 0.25] | 0 [0 to 0]

7. Secondary Outcome: Change of DCFPyL-PET/MRI Positive Lesions
Description: 18F-DCFPyL Positron Emission Tomography (PET)/MRI or -PET/CT positive sites that are positive for new or progressive metastatic disease by bone scan/CT at 6-months following SBRT.
Time Frame: 6 months
Population: Data was not collected for this outcome measure
Arm/Group | Observational (no SBRT) | SBRT
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Survival of Two Groups as Assessed by PSA Level
Description: The PSA levels in blood will be measured in units of nanograms per milliliter (ng/mL).
Time Frame: Baseline and 6 months
Population: Data was not collected
Arm/Group | SBRT | Observational (no SBRT)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Androgen Deprivation Therapy-free Survival
Description: Androgen Deprivation Therapy-free survival will be assessed using the number of participants deceased at 6 months.
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Observational (no SBRT) | SBRT
Number analyzed (Participants) | 18 | 36
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 6 months
Arm/Group | Observational (no SBRT) | SBRT
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/36
Other Adverse Events (participants affected / at risk) | 14/18 | 36/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational (no SBRT) (N=18) | SBRT (N=36)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 1 (1) — 6 month
Fatigue (General disorders) | 1 (1) | 1 (1) — 6 month
Anorexia (General disorders) | 1 (1) | 0 (0) — 6 month
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — 6 month
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) — 6 month
Depression (Psychiatric disorders) | 0 (0) | 1 (1) — 6 month
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — 6 month
Weight loss (General disorders) | 0 (0) | 1 (1) — 6 month
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — 6 month
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) — 6 month
Weight gain (General disorders) | 0 (0) | 1 (1) — 6 month
Dry mouth (General disorders) | 0 (0) | 1 (1) — 6 month
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) — 6 month
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — 6 month
Perineal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — 6 month
Insomnia (General disorders) | 0 (0) | 1 (1) — 6 month
Bladder infection (Renal and urinary disorders) | 0 (0) | 1 (1) — 6 month
Urinary Incontinence (Renal and urinary disorders) | 2 (2) | 2 (2) — 3 month
Bruising (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — 3 month
Fatigue (General disorders) | 1 (1) | 5 (5) — 3 month
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) — 3 month
Urinary Retention (Renal and urinary disorders) | 1 (1) | 1 (1) — 3 month
Localized Edema (General disorders) | 1 (1) | 2 (2) — 3 month
Depression (Psychiatric disorders) | 1 (1) | 0 (0) — 3 month
Tremor (General disorders) | 1 (1) | 0 (0) — 3 month
Pruritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — 3 month
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) — 3 month
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) — 3 month
Weight Loss (General disorders) | 0 (0) | 2 (2) — 3 month
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) — 3 month
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) — 3 month
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) — 3 month
Anemia (General disorders) | 0 (0) | 1 (1) — 3 month
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) — 3 month
Dizziness (General disorders) | 0 (0) | 1 (1) — 3 month
Dehydration (General disorders) | 0 (0) | 1 (1) — 3 month
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) — 3 month
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — 3 month
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — 3 month

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT02680587/Prot_SAP_000.pdf